CLINICAL TRIAL: NCT00421213
Title: Phase II Study of ZIO-101 in Advanced Blood and Bone Marrow Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGL2003
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Hematologic Neoplasms; Bone Marrow Neoplasms; Non-Hodgkin's Lymphoma
Keywords: APL; Lymphoma; T-cell Lymphoma; Peripheral T-cell Lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Bone Marrow Neoplasms; Lymphoma, Non-Hodgkin; Lymphoma; Lymphoma, T-Cell; Lymphoma, T-Cell, Peripheral | interventions — darinaparsin

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Darinaparsin

INTERVENTIONS:
Drug: Darinaparsin — 300mg/m2 of Darinaparsin given daily for five consecutive days to be repeated every 28 days for up to six months.
  Other Names: ZIO-101

SUMMARY:
The study of safety of a new organic arsenic compound in the treatment of hematological malignancies.

ELIGIBILITY:
Inclusion Criteria

1. Hodgkin's or non-Hodgkin's Lymphoma.
2. ≥ 1 prior therapy and currently requiring therapy.
3. Evaluable disease (defined by disease-specific criteria listed in Appendix 1)
4. ≥ 18 years of age.
5. ECOG performance score ≤ 2 (see Appendix 2).
6. Life-expectancy ≥ 2 months.
7. Written informed consent in compliance with ZIOPHARM policies and the Human Investigation Review Committee with jurisdiction over the site.
8. No anti-cancer therapy exception of hydroxyurea ≤ 3 weeks before Baseline (Day 1, Cycle 1).
9. The following clinical laboratory values < 2 weeks before Baseline:

   * Creatinine ≤ 2X upper limit of normal (ULN).
   * Total bilirubin ≤ 2X ULN.
   * Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 3X ULN.

Exclusion Criteria

1. New York Heart Association (NYHA) functional class ≥3 myocardial infarction (see Appendix ) within 6 months before Baseline or uncontrolled cardiac arrhythmia other than asymptomatic atrial fibrillation; a QTc ≥450 msec; or a ≥grade-2 atrioventricular (AV) block or left bundle branch block (LBBB).
2. Pregnant and/or lactating female. (Women of childbearing age must use effective contraception from Screening through the duration of study participation).
3. Uncontrolled infection.
4. Prior seizures ≥ grade-3 in CTC v.3 criteria.
5. Arsenic allergy.
6. Significant neuropathology, defined as grade > 2 per CTCAE Version 3.0.
7. Confusion or dementia.
8. Prior history of neurological deficits (e.g., stroke, dementia, ischemia) that has the potential to confound a post-dose neurological assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Response Rate | 6 months

SECONDARY OUTCOMES:
toxicities | 6 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Miami, Florida
  - Chicago, Illinois
  - Bethesda, Maryland
  - Fargo, North Dakota
  - Sioux Falls, South Dakota
  - Morgantown, West Virginia